CLINICAL TRIAL: NCT01239901
Title: Iron-mediated Vascular Disease in Sickle Cell Disease.
Brief Title: Iron Mediated Vascular Disease in Sickle Cell Anemia Patients
Status: Completed | Type: Observational
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, John C. Wood, Associate Professor of Pediatrics - Division of Cardiology, Children's Hospital Los Angeles
Other Study IDs: 1RC1HL099412-01 (NIH)
Record Dates: First submitted 2010-11-12; First posted 2010-11-15 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; sickle cell anemia; sickled cells; blood vessel; iron overload
MeSH Terms: conditions — Anemia, Sickle Cell; Iron Overload

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Red Blood Cells (RBCs), Peripheral Blood Mononuclear Cells (PBMCs), Plasma, Serum, and Urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this research study is to determine the frequency and severity of iron overload in patients with Sickle Cell Anemia and its relationship to blood vessel function. The investigators hypothesize that intermittent transfusions that these patients receive during hospitalizations produces significant iron overload and impairs blood vessel relaxation.

DETAILED DESCRIPTION:
Patients with sickle cell anemia often require blood transfusion as part of the treatment for their disease. Each teaspoon of transfused blood contains about 5 mg of iron and the levels of iron in sickle cell patients increase rapidly with each transfusion. While iron is necessary for many bodily functions, too much iron damages blood vessels, liver, hormone producing glands (pancreas, pituitary and thyroid) and the heart. It is important to know how iron damages blood vessels because most of the problems experienced by sickle cell anemia patients (stroke, kidney failure, pulmonary hypertension, heart disease) result from blood vessel damage. In this trial, iron in the liver, pancreas, and kidney will be measured noninvasively by MRI while vascular function will be measured by ultrasound and tissue Doppler. Patients will be recruited primarily from the greater Los Angeles area, although patients from greater distances will be allowed to participate.

ELIGIBILITY:
Inclusion Criteria:

* Age > 13 years
* Documented diagnosis of sickle cell anemia (SS, SC, Sß0, Sß+)
* Transfused no more than 8 times in a year.

Exclusion Criteria:

* Cardiac pacemaker, implantable neurostimulator or other MRI incompatible device.
* History of extreme claustrophobia in MRI machine or other reason for inability to do MRI without sedation.
* Inability to be positioned on the MRI table for sufficient time to complete the MRI exams.
* Any medical or psychological condition that, in the opinion of the local investigator, would make it unsafe or ill-advised for the subject to participate.
* Currently not receiving chronic transfusion therapy, defined as greater than 8 transfusions per year.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Our large and well-established sickle cell Center has strong ties to the SCD community in a large metropolitan area (Los Angeles), placing us in an ideal position to rapidly accrue sufficient subjects to study the prevalence of iron overload and determine the relation between directly measured iron loading, vascular responsiveness and clinically relevant biomarkers of vascular function.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2009-12; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Liver iron concentration (LIC), pancreas R2*, and kidney R2*, measured by MRI | 15 min MRI done completed during one time study visit
  Liver iron concentration (LIC) will be used as a surrogate for total body iron, pancreatic iron represents a surrogate for extravascular iron deposition, and renal iron as a surrogate for chronic intravascular hemolysis. In addition, labile plasma iron will be measured in blood plasma.

SECONDARY OUTCOMES:
Vascular function. | Scheduled during one time study visit
  Measurements will be done through several procedures: Ultrasound of artery in upper arm, Ultrasound of artery in neck, and blood tests of ascorbate and hydrobiopterins.

CONTACTS AND LOCATIONS:
Overall Officials: John C Wood, MD, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ballas SK. Iron overload is a determinant of morbidity and mortality in adult patients with sickle cell disease. Semin Hematol. 2001 Jan;38(1 Suppl 1):30-6. doi: 10.1016/s0037-1963(01)90058-7. PMID 11206959
- [Background] Cheung YF, Chan GC, Ha SY. Effect of deferasirox (ICL670) on arterial function in patients with beta-thalassaemia major. Br J Haematol. 2008 May;141(5):728-33. doi: 10.1111/j.1365-2141.2008.07092.x. Epub 2008 Mar 3. PMID 18318756
- [Background] Borgna-Pignatti C, Rugolotto S, De Stefano P, Zhao H, Cappellini MD, Del Vecchio GC, Romeo MA, Forni GL, Gamberini MR, Ghilardi R, Piga A, Cnaan A. Survival and complications in patients with thalassemia major treated with transfusion and deferoxamine. Haematologica. 2004 Oct;89(10):1187-93. PMID 15477202
- [Background] Pakbaz Z, Fischer R, Fung E, Nielsen P, Harmatz P, Vichinsky E. Serum ferritin underestimates liver iron concentration in transfusion independent thalassemia patients as compared to regularly transfused thalassemia and sickle cell patients. Pediatr Blood Cancer. 2007 Sep;49(3):329-32. doi: 10.1002/pbc.21275. PMID 17554789
- [Background] Schein A, Enriquez C, Coates TD, Wood JC. Magnetic resonance detection of kidney iron deposition in sickle cell disease: a marker of chronic hemolysis. J Magn Reson Imaging. 2008 Sep;28(3):698-704. doi: 10.1002/jmri.21490. PMID 18777554
- [Background] Wood JC, Enriquez C, Ghugre N, Tyzka JM, Carson S, Nelson MD, Coates TD. MRI R2 and R2* mapping accurately estimates hepatic iron concentration in transfusion-dependent thalassemia and sickle cell disease patients. Blood. 2005 Aug 15;106(4):1460-5. doi: 10.1182/blood-2004-10-3982. Epub 2005 Apr 28. PMID 15860670
- [Background] Wood JC, Enriquez C, Ghugre N, Otto-Duessel M, Aguilar M, Nelson MD, Moats R, Coates TD. Physiology and pathophysiology of iron cardiomyopathy in thalassemia. Ann N Y Acad Sci. 2005;1054:386-95. doi: 10.1196/annals.1345.047. PMID 16339687
- [Background] Ganz T. Molecular control of iron transport. J Am Soc Nephrol. 2007 Feb;18(2):394-400. doi: 10.1681/ASN.2006070802. Epub 2007 Jan 17. PMID 17229910
- [Background] Oudit GY, Trivieri MG, Khaper N, Liu PP, Backx PH. Role of L-type Ca2+ channels in iron transport and iron-overload cardiomyopathy. J Mol Med (Berl). 2006 May;84(5):349-64. doi: 10.1007/s00109-005-0029-x. Epub 2006 Apr 8. PMID 16604332
- [Background] Walter PB, Fung EB, Killilea DW, Jiang Q, Hudes M, Madden J, Porter J, Evans P, Vichinsky E, Harmatz P. Oxidative stress and inflammation in iron-overloaded patients with beta-thalassaemia or sickle cell disease. Br J Haematol. 2006 Oct;135(2):254-63. doi: 10.1111/j.1365-2141.2006.06277.x. PMID 17010049
- [Background] Kato GJ, Gladwin MT. Evolution of novel small-molecule therapeutics targeting sickle cell vasculopathy. JAMA. 2008 Dec 10;300(22):2638-46. doi: 10.1001/jama.2008.598. PMID 19066384
- [Background] Vanhoutte PM, Shimokawa H, Tang EH, Feletou M. Endothelial dysfunction and vascular disease. Acta Physiol (Oxf). 2009 Jun;196(2):193-222. doi: 10.1111/j.1748-1716.2009.01964.x. Epub 2009 Feb 10. PMID 19220204
- [Background] Morris CR, Kato GJ, Poljakovic M, Wang X, Blackwelder WC, Sachdev V, Hazen SL, Vichinsky EP, Morris SM Jr, Gladwin MT. Dysregulated arginine metabolism, hemolysis-associated pulmonary hypertension, and mortality in sickle cell disease. JAMA. 2005 Jul 6;294(1):81-90. doi: 10.1001/jama.294.1.81. PMID 15998894
- [Background] Werner ER, Gorren AC, Heller R, Werner-Felmayer G, Mayer B. Tetrahydrobiopterin and nitric oxide: mechanistic and pharmacological aspects. Exp Biol Med (Maywood). 2003 Dec;228(11):1291-302. doi: 10.1177/153537020322801108. PMID 14681545
- [Background] Valenti L, Fracanzani AL, Dongiovanni P, Bugianesi E, Marchesini G, Manzini P, Vanni E, Fargion S. Iron depletion by phlebotomy improves insulin resistance in patients with nonalcoholic fatty liver disease and hyperferritinemia: evidence from a case-control study. Am J Gastroenterol. 2007 Jun;102(6):1251-8. doi: 10.1111/j.1572-0241.2007.01192.x. Epub 2007 Mar 27. PMID 17391316
- [Background] Tanner MA, Galanello R, Dessi C, Smith GC, Westwood MA, Agus A, Roughton M, Assomull R, Nair SV, Walker JM, Pennell DJ. A randomized, placebo-controlled, double-blind trial of the effect of combined therapy with deferoxamine and deferiprone on myocardial iron in thalassemia major using cardiovascular magnetic resonance. Circulation. 2007 Apr 10;115(14):1876-84. doi: 10.1161/CIRCULATIONAHA.106.648790. Epub 2007 Mar 19. PMID 17372174
- [Background] Castro O, Haddy TB. Improved survival of iron-deficient patients with sickle erythrocytes. N Engl J Med. 1983 Mar 3;308(9):527. No abstract available. PMID 6823275
- [Background] Gladwin MT, Sachdev V, Jison ML, Shizukuda Y, Plehn JF, Minter K, Brown B, Coles WA, Nichols JS, Ernst I, Hunter LA, Blackwelder WC, Schechter AN, Rodgers GP, Castro O, Ognibene FP. Pulmonary hypertension as a risk factor for death in patients with sickle cell disease. N Engl J Med. 2004 Feb 26;350(9):886-95. doi: 10.1056/NEJMoa035477. PMID 14985486
- [Background] de Montalembert M, Aggoun Y, Niakate A, Szezepanski I, Bonnet D. Endothelial-dependent vasodilation is impaired in children with sickle cell disease. Haematologica. 2007 Dec;92(12):1709-10. doi: 10.3324/haematol.11253. PMID 18055999
- [Background] Belhassen L, Pelle G, Sediame S, Bachir D, Carville C, Bucherer C, Lacombe C, Galacteros F, Adnot S. Endothelial dysfunction in patients with sickle cell disease is related to selective impairment of shear stress-mediated vasodilation. Blood. 2001 Mar 15;97(6):1584-9. doi: 10.1182/blood.v97.6.1584. PMID 11238095
- [Background] Takeda M, Yamashita T, Shinohara M, Sasaki N, Takaya T, Nakajima K, Inoue N, Masano T, Tawa H, Satomi-Kobayashi S, Toh R, Sugiyama D, Nishimura K, Yokoyama M, Hirata K, Kawashima S. Plasma tetrahydrobiopterin/dihydrobiopterin ratio: a possible marker of endothelial dysfunction. Circ J. 2009 May;73(5):955-62. doi: 10.1253/circj.cj-08-0850. Epub 2009 Mar 18. PMID 19293532
- [Background] Gonzalez J, Wood JC, Dorey FJ, Wren TA, Gilsanz V. Reproducibility of carotid intima-media thickness measurements in young adults. Radiology. 2008 May;247(2):465-71. doi: 10.1148/radiol.2472070691. Epub 2008 Mar 18. PMID 18349312
- [Background] Cheung YF, Chow PC, Chan GC, Ha SY. Carotid intima-media thickness is increased and related to arterial stiffening in patients with beta-thalassaemia major. Br J Haematol. 2006 Dec;135(5):732-4. doi: 10.1111/j.1365-2141.2006.06349.x. PMID 17107355
- [Background] Kato GJ, McGowan V, Machado RF, Little JA, Taylor J 6th, Morris CR, Nichols JS, Wang X, Poljakovic M, Morris SM Jr, Gladwin MT. Lactate dehydrogenase as a biomarker of hemolysis-associated nitric oxide resistance, priapism, leg ulceration, pulmonary hypertension, and death in patients with sickle cell disease. Blood. 2006 Mar 15;107(6):2279-85. doi: 10.1182/blood-2005-06-2373. Epub 2005 Nov 15. PMID 16291595
- [Background] Morris CR, Suh JH, Hagar W, Larkin S, Bland DA, Steinberg MH, Vichinsky EP, Shigenaga M, Ames B, Kuypers FA, Klings ES. Erythrocyte glutamine depletion, altered redox environment, and pulmonary hypertension in sickle cell disease. Blood. 2008 Jan 1;111(1):402-10. doi: 10.1182/blood-2007-04-081703. Epub 2007 Sep 11. PMID 17848621